CLINICAL TRIAL: NCT05713006
Title: A Phase I/II Open-label Clinical Trial to Evaluate the Pharmacokinetics of Alectinib With Sequential Dose Escalation in Patients Diagnosed With ALK-rearranged Advanced Non-small Cell Lung Cancer.
Brief Title: Alectinib Pharmacokinetic in Patients With NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of the Thoracic Oncology Unit and Personalized Medicine Laboratory, Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022/023/ICI_CEI/1583/21_V.2
Record Dates: First submitted 2023-01-04; First posted 2023-02-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB; ALK Gene Mutation
Keywords: alectinib; positive-ALK; non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Intervention Model Description: Patients (≥18 years), both sex, clinical stage IIIB and IV, ALK-rearranged NSCLC treated by Thoracic Oncology Department at Instituto Nacional de Cancerología (INCan).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Alectinib escalation dose (Experimental): Alecensa 150 mg Roche
  Interventions: Drug: Alectinib Oral Product

INTERVENTIONS:
Drug: Alectinib Oral Product — Alectinib is administered with a sequential dose escalation every 21 days from 300 to 600mg twice daily in the phase 1 portion. In phase 2, patients received an investigator-chosen dose based on the PK analysis.
  Other Names: Alecensa 150 mg Roche

SUMMARY:
This interventional study aims to determine the pharmacokinetics of orally administered alectinib with dose escalation from 300 mg to 600 mg twice daily in Mexican patients with advanced ALK-positive NSCLC.

The main question it aims to answer is: what will be the peak plasma concentrations of alectinib following sequential dose escalation (300, 450, and 600 mg BID) over nine weeks of pharmacokinetic evaluation (phase I) in Mexican patients with advanced ALK-rearranged NSCLC?

In phase I (on days 0, 21, and 42), oral alectinib will be administered twice per day (BID) to patients with ALK-positive NSCLC; starting with 300 mg BID in 21-day cycles and dose escalation in 150 mg increments until 600 mg BID. Blood samples will be taken before and after administration of each dose (on days 1, 22, and 43). The primary endopoints in phase I will be dose-limiting toxicity (DLT) and PK parameters (Cmax. maximum plasma concentration; Tmax: time to reach maximum concentration: AUC 1-12: area under plasma ocncentrations-time curve steady-state concentration). At the end of the last blood collection (at day 43), the evaluation of each cycle will be at 600 mg, and the participant will be discharged to continue their treatment on an outpatient basis. Phase one will finish on day 63 of the study.

In phase II, the chosen BID dose based on the phase I portion will be administrated until disease progression, development of unacceptable side effects, or withdrawal of consent. The primary endpoint in phase 2 is the overall response rate (ORR) per RECIST V.1.1.

DETAILED DESCRIPTION:
Alectinib will be administrated under fast conditions.

The primary endpoint of the phase II part was ORR. Other secondary endpoints in phase II are progression-free survival (PFS), overall survival (OS), intracranial response (ICR), and duration of response (DOR).

Exploratory endpoints in this follow-up analysis included the evaluation of the correlation between tumor shrinkage and PFS and chosen dose to relieve cancer symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* ≥ 18 years old
* Pathologically confirmed diagnosis of NSCLC
* Stage IIIB - IV by the American Joint Committee of Cancer Version 8.
* Recurrent disease (at least 180 days from curative intent treatment)
* ALK rearrangements tested by FDA-approved tests (IHQ or FISH)
* Karnofsky PS scale ≥ 70%
* Having received first-line treatment with anti-ALK inhibitors and one previous line of platinum-based chemotherapy.
* Measurable disease as referred by RECIST version 1.1
* Symptomatic brain metastases could receive prior treatment with radiotherapy or surgery for at least two weeks before treatment initiation.
* Asymptomatic brain metastases could not receive local therapy before study inclusion.
* Negative highly sensitive pregnancy test (serum or urine) within 72 days before first dose intervention.
* Sexually active patients should use a contraceptive method with a failure rate of less than 1% per year.
* Signed written informed consent
* Adequate organ function (hematological, liver, and renal function)
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Carcinomatous meningitis confirmed by a positive CRL cytology or highly suspicious brain MRI.
* Previous malignancies except for any carcinoma in-situ
* Treatment with other anti-cancer therapy
* Participating in other clinical trials in the former four weeks
* Any other serious condition or uncontrolled active infection, altered mental status, or psychiatric condition that, in the investigator´s opinion, would limit the ability of an individual to meet the requirements of the study or which affects the interpretability of the results.
* Active hepatitis virus infection (any serotype) or chronic infection with a potential risk of reactivation evaluated through a serological panel.
* Active HIV infection.
* Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
AUC | Amount of drug concentration between 0 to 12 hours after first drug administration
  The area under the curve (AUC). Pharmacokinetic behavior of the initial alectinib for each given dose (300, 450 and 600 mg).
Cmax | From baseline control pre-dose, 0.50, 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00 and 11.90 hours
  Highest concentration of drug in blood (Serum) for each given dose (300, 450 and 600 mg).
Cmin | From baseline control pre-dose, 0.50, 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00 and 11.90 hours
  Lowest concentration of drug in blood (Serum) for each given dose (300, 450 and 600 mg).
Tmax | From first dose administration through the following 12 hours (day 1)
  Time in witch Cmax is reached in each dose of the drug (300,450 and 600 mg)
ORR | From first dose administration up to disease progression by CT scan every 6 weeks, through study completion.
  overall response rate is measured in phase two
Steady state | For phase two: between 2 and 4 months of treatment with investigators chosen dose.
  The amount of drug in the plasma has built up to a therapeutically effective concentration level, and as long as regular doses are administered to balance the amount of drug being cleared, the drug will continue to be active.

SECONDARY OUTCOMES:
Adverse events | From date of first dose administration through 9 weeks.
  Tolerance during drug escalation doses (300, 450, and 600 mg) in the phase one portion based on the PK analysis.
Drug toxicity | From date of starting phase 2 portion until the date of first documented progression date or death from any cause, whichever comes first, assessed up to 60 months.
  Adverse events under alectinib Administration a the chosen dose are measured in the phase two portion.
PFS | From date of first dose administration until the date of first documented progression date or death from any cause, whichever comes first, assessed up to 100 months.
  Progression-free survival
OS | From date of first dose administration until the date of documented death from any cause or last follow-up, whichever comes first, assessed up to 120 months.
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta Rodriguez, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Thoracic Oncology Unit and Personalized Medicine Laboratory, Instituto Nacional de Cancerología, Mexico City, Mexico

REFERENCES:
- [Background] Morcos PN, Nueesch E, Jaminion F, Guerini E, Hsu JC, Bordogna W, Balas B, Mercier F. Exposure-response analysis of alectinib in crizotinib-resistant ALK-positive non-small cell lung cancer. Cancer Chemother Pharmacol. 2018 Jul;82(1):129-138. doi: 10.1007/s00280-018-3597-5. Epub 2018 May 10. PMID 29748847
- [Background] Sivignon M, Monnier R, Tehard B, Roze S. Cost-effectiveness of alectinib compared to crizotinib for the treatment of first-line ALK+ advanced non-small-cell lung cancer in France. PLoS One. 2020 Jan 16;15(1):e0226196. doi: 10.1371/journal.pone.0226196. eCollection 2020. PMID 31945065
- [Background] Carlson JJ, Suh K, Orfanos P, Wong W. Cost Effectiveness of Alectinib vs. Crizotinib in First-Line Anaplastic Lymphoma Kinase-Positive Advanced Non-Small-Cell Lung Cancer. Pharmacoeconomics. 2018 Apr;36(4):495-504. doi: 10.1007/s40273-018-0625-6. PMID 29488070
- [Background] Hida T, Nokihara H, Kondo M, Kim YH, Azuma K, Seto T, Takiguchi Y, Nishio M, Yoshioka H, Imamura F, Hotta K, Watanabe S, Goto K, Satouchi M, Kozuki T, Shukuya T, Nakagawa K, Mitsudomi T, Yamamoto N, Asakawa T, Asabe R, Tanaka T, Tamura T. Alectinib versus crizotinib in patients with ALK-positive non-small-cell lung cancer (J-ALEX): an open-label, randomised phase 3 trial. Lancet. 2017 Jul 1;390(10089):29-39. doi: 10.1016/S0140-6736(17)30565-2. Epub 2017 May 10. PMID 28501140
- [Background] Peters S, Camidge DR, Shaw AT, Gadgeel S, Ahn JS, Kim DW, Ou SI, Perol M, Dziadziuszko R, Rosell R, Zeaiter A, Mitry E, Golding S, Balas B, Noe J, Morcos PN, Mok T; ALEX Trial Investigators. Alectinib versus Crizotinib in Untreated ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Aug 31;377(9):829-838. doi: 10.1056/NEJMoa1704795. Epub 2017 Jun 6. PMID 28586279